CLINICAL TRIAL: NCT03805841
Title: Phase 2 Study - Evaluate the Clinical Activity of Tarloxotinib in Patients With Non-Small Cell Lung Cancer That Harbors an EGFR Exon 20 Insertion or HER2-Activating Mutation and Other Advanced Solid Tumors With NRG1/ERBB Family Gene Fusions
Brief Title: Study of Tarloxotinib in Pts With NSCLC (EGFR Exon 20 Insertion, HER2-activating Mutations) & Other Solid Tumors With NRG1/ERBB Gene Fusions
Acronym: RAIN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: enrollment pause
Sponsor: Rain Oncology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAIN-701
Record Dates: First submitted 2019-01-11; First posted 2019-01-16 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-04

CONDITIONS: NSCLC, Stage IV; NSCLC Stage IIIB; NSCLC, Stage IIIC; NSCLC, Recurrent; EGFR Exon 20 Insertion Mutation; HER2-activating Mutation; ERBB Fusion; NRG1 Fusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): tarloxotinib bromide
  Interventions: Drug: tarloxotinib bromide

INTERVENTIONS:
Drug: tarloxotinib bromide — weekly intravenous infusion
  Other Names: Tarlox; tarloxotinib

SUMMARY:
Open-label, Phase 2, single treatment arm, 3 cohorts

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically and/or cytologically confirmed primary diagnosis of NSCLC, Stage IV, Stage IIIB or IIIC not amenable to definitive curative intent therapy, or recurrent disease after prior diagnosis of Stage I-III disease. Cohort C locally advanced or metastatic solid tumor.
* Progression of disease on or after a platinum-based chemotherapy regimen (Cohorts A and B) or after standard of care (Cohort C)
* EGFR exon 20 insertion mutation (Cohort A) or HER2 activating mutation (Cohort B) or NRG1 or ERBB family gene fusions (Cohort C)
* Measurable disease according to RECIST v.1.1
* ECOG performance status of 0 or 1
* Serum creatinine ≤ 1.5 x ULN (or calculated creatinine clearance ≥ 60 mL/min using Cockcroft Gault equation)
* Total bilirubin: ≤ 1.5 x ULN or ≤ 3 x ULN in the presence of liver metastases
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN, or ≤ 5 x ULN, in the presence of liver metastases
* Absolute neutrophil count (ANC) ≥ 1,500 cells/μL
* Hemoglobin ≥ 9 g/dL or 5.6 mmol/L
* Platelet count ≥ 100,000/μL
* No evidence of second or third degree atrioventricular block
* No clinically significant arrhythmia (i.e.; pauses of > 4 seconds, VT of any duration, SVT > 4 beats/minute)
* QRS interval ≤ 110 ms
* QTcF interval of < 450 ms
* PR interval ≤ 200 ms
* Adequate pretreatment tumor sample (125 µm of FFPE block or at least 8 prepared slides)

Key Exclusion Criteria:

* Another known activating oncogene driver mutation
* (Cohorts A and B Only) Previously received anti EGFR or anti HER2 tyrosine kinase inhibitors
* (Cohorts A and B Only) Previously received anti EGFR or anti HER2 monoclonal antibodies or EGFR or HER2 antibody drug conjugates
* Investigational therapy administered within the 28 days or 5 half lives
* Chemotherapy or radiation within 14 days prior to Cycle 1 Day 1
* Immunotherapy within 21 days
* Clinically active or symptomatic interstitial lung disease (ILD) or interstitial pneumonitis, or a history of clinically significant ILD or radiation pneumonitis
* Untreated and/or symptomatic CNS malignancies (primary or metastatic);
* Receiving medication that prolongs QT interval, with a risk of causing Torsade de Pointes (TdP)
* Personal or familial history of Long QT Syndrome
* NYHA class III or IV or LVEF < 55%
* Myocardial infarction, severe or unstable angina within 6 months
* History of TdP, ventricular arrhythmia
* Significant thrombotic or embolic events within 3 months
* Uncontrolled or severe cardiovascular disease
* Concurrent malignancy expected to require treatment within 2 years or interfere with study outcomes
* History of severe allergic reactions or hypersensitivity to compounds of similar chemical or biologic composition as tarloxotinib
* Known HIV infection or active Hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen V Liu, MD, Principal Investigator — Georgetown University
Locations (14):
- United States (11):
  - RAIN-701 Study Site, Irvine, California
  - Pacific Shores Medical Group, Long Beach, California
  - University of California San Francisco, Helen Diller Cancer Center, San Francisco, California
  - RAIN-701 Study Site, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Comprehensive Care and Research Center, Atlanta, Newnan, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Providence Cancer Institute, Portland, Oregon
  - RAIN-701 Study Site, Pittsburgh, Pennsylvania
  - RAIN-701 Study Site, Seattle, Washington
- RAIN-701 Study Site, Toronto, Ontario, Canada
- Hong Kong (2):
  - RAIN-701 Study Site, Hong Kong
  - Hong Kong United Oncology Center, Kowloon

IPD SHARING:
Plan to Share IPD: No
No Plan

REFERENCES:
- [Derived] Ye L, Chen X, Zhou F. EGFR-mutant NSCLC: emerging novel drugs. Curr Opin Oncol. 2021 Jan;33(1):87-94. doi: 10.1097/CCO.0000000000000701. PMID 33122578

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (N=11): Previously treated advanced/metastatic non-small cell lung cancer (NSCLC) who have a tumor harboring an EGFR exon 20 insertion.
  Subjects received taroxontinib 150 mg/m2 administered as a weekly 1-hour IV infusion on Days 1, 8, 15, and 22 of each 28-day cycle until disease progression or unacceptable toxicity.
- Cohort B (N=22): Previously treated advanced/metastatic non-small cell lung cancer (NSCLC) who have a tumor harboring a HER2-activating mutation (including HER2 exon 20 insertions) who have not received prior HER2-directed therapy.
  Subjects received taroxontinib 150 mg/m2 administered as a weekly 1-hour IV infusion on Days 1, 8, 15, and 22 of each 28-day cycle until disease progression or unacceptable toxicity
- Cohort C (N=8): Previously treated advanced solid tumors harboring NRG1 or ERBB/HER-family gene fusions.
  Subjects received taroxontinib 150 mg/m2 administered as a weekly 1-hour IV infusion on Days 1, 8, 15, and 22 of each 28-day cycle until disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Cohort A (N=11) | Cohort B (N=22) | Cohort C (N=8)
Started | 11 | 22 | 8
Completed | 6 | 12 | 5
Not Completed | 5 | 10 | 3
Not completed — Clinical Progression | 2 | 0 | 0
Not completed — Death | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 0
Not completed — Progressive disease according to RECIST 1.1 at any time during the study | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A (N=11): Previously treated advanced/metastatic non-small cell lung cancer (NSCLC) who have a tumor harboring an EGFR exon 20 insertion
- Cohort B (N=22): Previously treated advanced/metastatic non-small cell lung cancer (NSCLC) who have a tumor harboring a HER2-activating mutation (including HER2 exon 20 insertions) who have not received prior HER2-directed therapy
- Cohort C (N=8): Previously treated advanced solid tumors harboring NRG1 or ERBB/HER-family gene fusions
- Total: Total of all reporting groups
Arm/Group | Cohort A (N=11) | Cohort B (N=22) | Cohort C (N=8) | Total
Number analyzed (Participants) | 11 | 22 | 8 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 17 | 6 | 29
  >=65 years | 5 | 5 | 2 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 5 | 23
  Male | 4 | 11 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 4
  Not Hispanic or Latino | 10 | 19 | 7 | 36
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 4 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 5 | 13 | 4 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5
Smoking Status, n(%) [Count of Participants; unit: Participants]
  Non-Smoker | 9 | 17 | 5 | 31
  Former Smoker | 2 | 3 | 2 | 7
  Current Smoker | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: ORR
Description: The primary objective of this study is to evaluate the objective response rate (ORR) of tarloxotinib according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for tumors assessed by CT or MRI: Complete Response (CR) - Disappearance of all target lesions and reduction in the short axis measurement of all pathologic lymph nodes to ≤10 mm. Partial Response (PR) - ≥30% decrease in the sum of the longest diameter of the target lesions compared with baseline.
  The overall response rate in each cohort will be estimated as the number of subjects with a confirmed objective response (CR or PR) divided by the number of enrolled subjects in each respective cohort.
Time Frame: Through study completion, an average of 10 months.
Population: The Primary Analysis Set, referred to as the Safety Population in the protocol, is defined as all subjects who subjects who received at least 1 dose of tarloxotinib. The Primary Analysis Set will be the analysis population for the safety and efficacy analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (N=11) | Cohort B (N=22) | Cohort C (N=8)
Number analyzed (Participants) | 11 | 22 | 8
percentage of participants | 0 [0.00 to 28.49] | 13.6 [2.91 to 34.91] | 0 [0.00 to 36.94]

ADVERSE EVENTS:
Time Frame: From time of first dose, through 30 days after last dose, up to 12 months.
Description: Safety was assessed by repeated clinical evaluations including adverse events (AEs), suspected adverse reactions, unexpected events, serious AEs (SAEs), serious unexpected suspected adverse reactions, vital signs, physical examination, ECGs, clinical laboratory tests (serum chemistry, hematology, and urinalysis ).
Arm/Group | Cohort A (N=11) | Cohort B (N=22) | Cohort C (N=8)
All-Cause Mortality (participants affected / at risk) | 5/11 | 4/22 | 1/8
Serious Adverse Events (participants affected / at risk) | 4/11 | 9/22 | 3/8
Other Adverse Events (participants affected / at risk) | 11/11 | 22/22 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=11) (N=11) | Cohort B (N=22) (N=22) | Cohort C (N=8) (N=8)
Lung infection (Infections and infestations) | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hemmorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=11) (N=11) | Cohort B (N=22) (N=22) | Cohort C (N=8) (N=8)
Rash (Skin and subcutaneous tissue disorders) | 5 | 9 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 7 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 8 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 6 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 10 | 19 | 6
Alanine aminotransferase increased (Investigations) | 2 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 1
Lymphocyte count decreased (Investigations) | 0 | 2 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 2 | 0
Lymphocyte count increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 5
Nausea (Gastrointestinal disorders) | 3 | 5 | 2
Constipation (Gastrointestinal disorders) | 2 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2
Paraesthesia oral (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Tongue discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 3 | 3
Oedema peripheral (General disorders) | 1 | 2 | 1
Pyrexia (General disorders) | 2 | 2 | 0
Asthenia (General disorders) | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 2 | 0
Application site pruritus (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Infusion site erythema (General disorders) | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Tenderness (General disorders) | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Arthralgia (Metabolism and nutrition disorders) | 0 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bladder irritation (Renal and urinary disorders) | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0
Flushing (Vascular disorders) | 1 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Eye disorder (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-10-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT03805841/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03805841/SAP_001.pdf